CLINICAL TRIAL: NCT07156253
Title: A Phase Ib Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of SYN818 With Olaparib in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of SYN818 With Olaparib for the Treatment of Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou SynRx Therapeutics Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYN-818-102
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Solid Tumor; Ovarian Cancer; Breast Cancer; BRCA 1 /2 and / or HRD; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis; Ovarian Neoplasms; Breast Neoplasms; Kenny-Caffey syndrome, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYN818 combination with Olaparib (Experimental)
  Interventions: Drug: SYN818 and Olaparib will be administered

INTERVENTIONS:
Drug: SYN818 and Olaparib will be administered — Patients will orally receive SYN818 and Olaparib

SUMMARY:
This interventional study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of SYN818 with Olaparib in adult patients with locally advanced or metastatic solid tumors

DETAILED DESCRIPTION:
This study is a Phase Ib, open-label, multicentre study of SYN818 with Olaparib administered orally in patients with locally advanced or metastatic solid tumors harboring mutations in BRCA and/or defects in the homologous recombination repair (HRR) pathway

ELIGIBILITY:
Inclusion Criteria:

* Having signed the written Informed Consent Form (ICF);
* Male or female aged ≥18 years;
* Life expectancy ≥12 weeks;
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 or 1;
* Participant has a histologically confirmed diagnosis of advanced or metastatic solid tumor and has exhausted all standard-of-care treatment options, with documented BRCA mutations and/or homologous recombination repair deficiency (Part 1).
* Participant has histologically or cytologically confirmed locally advanced or metastatic epithelial ovarian cancer or HER2-negative breast cancer, with documented BRCA mutations and/or homologous recombination repair deficiency (Part 2).
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
* No serious hematological, cardiopulmonary, or liver or kidney diseases other than the primary disease;
* Adequate organ function and bone marrow function.

Exclusion Criteria:

* Previous or current use of DNA Polymerase Theta (POLQ) inhibitors;
* Current or previous other malignancy unless treated radically and with no evidence of recurrence or metastasis within the past 5 years;
* Central nervous system (CNS) metastasis or meningeal metastasis with clinical symptoms, or other evidence indicating that CNS metastasis or meningeal metastasis has not been adequately controlled;
* Patients with Myelodysplastic syndrome (MDS)/Acute myeloid leukemia (AML) or with features suggestive of MDS/AML;
* Dysphagia or refractory nausea and vomiting, malabsorption, extracorporeal biliary shunts, or gastrointestinal disorders that affect drug absorption, e.g., Crohn's disease, ulcerative colitis, or short bowel syndrome, or other malabsorption conditions;
* Treatment with an anti-cancer small molecule within 5 half-lives (t1/2), or 2 weeks, whichever is shorter;
* History of use within 2 weeks prior to the first dose of the study treatment and need to use protocol-prohibited potent inhibitors or potent inducers of cytochrome P450 (CYP) 3A4/BCRP/P-gp during the study;
* Serious systemic diseases or laboratory abnormalities or other conditions that, at the Investigator's discretion, will make it unsuitable for the patient to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-08-26 (Estimated); Primary Completion 2028-08-25 (Estimated); Study Completion 2029-02-25 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 3 years
  MTD is defined as the maximum dose level at which ≤1 patient have dose limiting toxicities (DLTs) during the DLT observation period, and it should be determined with 6 evaluable patients.
Number of participants with Dose Limiting Toxicities (DLTs) | From first dose of study treatment until the end of Cycle 1 (each cycle is 21-days)
  Severity of adverse events as assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Number of participants experiencing adverse events (AEs)/serious adverse events (SAEs) | From time of information consent to 30 days post last dose, up to 3 years
  Number of participants with incidence of adverse events and with serious adverse events including changes from baseline in laboratory parameters, vital signs, Electrocardiogram (ECG), and physical examination, etc.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK Peak Plasma Concentration (Cmax) of the SYN818 and Olaparib combination therapy
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK Time to Peak drug Concentration (Tmax) of the SYN818 and Olaparib combination therapy
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK Area under the plasma concentration versus time curve (AUC) of the combination therapy of SYN818 and Olaparib
Pharmacokinetic (PK) parameters | Up to 3 years
  To characterize the PK profile of the combination therapy of SYN818 and Olaparib by measuring elimination half-life (t1/2)
Objective Response Rate (ORR) | Up to 3 years
  ORR is defined as proportion of patients who achieved complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 recorded from first investigational product treatment until disease progression or death due to any cause. The confirmation of response for patients who has PR or CR at first time should be performed by at least 4 weeks. For castration-resistant prostate cancer (CRPC) patients, bone lesion will be assessed according to Prostate Cancer Working Group 3 (PCWG3) criteria.
Duration of Response (DoR) and Time to Response (TTR) | Up to 3 years
  DOR is defined, for patients with an objective response, as the time from first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or death due to any cause.
Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the time from the first study treatment to the date of the first documentation of objective progression of disease (PD) or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- FuDan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No